CLINICAL TRIAL: NCT02770651
Title: LAte Stent Strut APPosition and COverage After Drug-Eluting Stent ImplantaTIOn by Optical Coherence Tomography in PatieNts With Acute Myocardial Infarction II(APPOSITION-AMI II)
Brief Title: Late Stent Strut Apposition and Coverage After Drug-Eluting Stent Implantation by OCT in Patients With AMI
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Seung-Ho Hur, Professor of Internal Medicine, Keimyung University Dongsan Medical Center
Other Study IDs: 2016-01-030; APPOSITION-AMI II (Other: Keimyung University Dongsan Medical Center)
Record Dates: First submitted 2016-05-01; First posted 2016-05-12 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Arterial Occlusive Diseases; Arteriosclerosis; Cardiovascular Diseases; Heart Diseases; Vascular Diseases
Keywords: optical coherence tomography; everolimus-eluting stent; zotarolimus-eluting stent
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Arterial Occlusive Diseases; Arteriosclerosis; Cardiovascular Diseases; Heart Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Optical Coherence Tomography: To evaluate the incidence of late incomplete stent apposition (ISA) and un-coverage by optical coherence tomography (OCT) following everolimus-eluting stent (EES) with bioabsorbable polymerversus zotarolimus-eluting stent (ZES) with permanent polymer implantation in patients with AMI at 12 months.
  Interventions: Device: Everolimus-Eluting stent; Device: Zotarolimus-Eluting stent

INTERVENTIONS:
Device: Everolimus-Eluting stent — Everolimus-Eluting stent with bioabsorbable polymer
  Other Names: Synergy™
Device: Zotarolimus-Eluting stent — Zotarolimus-Eluting stent with permanent polymer
  Other Names: Resolute Onyx™

SUMMARY:
The purpose of this study is to evaluate the incidence of late incomplete stent apposition (ISA) and un-coverage by optical coherence tomography (OCT) following everolimus-eluting stent (EES) with bioabsorbable polymer (SYNERGY™, Boston Scientific,Nattick, MA, USA) versus zotarolimus-eluting stent (ZES) with permanent polymer(Resolute Onyx™, Medtronic, Santa Rosa, CA, USA) implantation in patients with AMI at 12 months.

DETAILED DESCRIPTION:
It has been known that persistence of polymer may affect the late/very late safety and efficacy of drug eluting stent (DES) although polymer provides a reservoir for programmed drug release. Newer durable polymers may have enhanced biocompatibility and seem to be associated with improved clinical outcomes. However, they have still been incriminated in the occurrence of inflammation, neo-atherosclerosis, and thrombosis. Therefore, the investigators will evaluate the vascular tissue reaction after different kinds of DES implantation under the high thrombogenic circumstance of acute myocardial infarction (AMI).

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction including ST-segment elevation myocardial infarction (STEMI) or non ST-segment elevation myocardial infarction (NSTEMI) treated with PCI
* Patient ≥ 18 years of age
* Patient judged suitable to receive anti-platelet drugs of ASA and ticagrelor for at least 12 months after the procedure
* The patient or guardian agrees to the study protocol and the schedule of clinical and angiographic, OCT follow up and provides informed consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.
* culprit lesion

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to any of the following medications: heparin, abciximab, aspirin, ticagrelor, everolimus, zotarolimus, polymer, platinum chromium, cobalt chromium, contrast media
* Female of childbearing potential unless a pregnancy test is negative or who possibly plan to become pregnant any time after enrollment
* Cardiogenic shock
* Patient with left ventricular ejection fraction <30%
* Patient with left main disease
* Patient with In-stent restenosis (ISR) at target vessel (either bare metal stent or DES, non-target vessel ISR is permitted)
* Patient with impaired renal function (creatinine >2.0mg/dL)
* Patient with inadequate OCT images quality due to severe calcification, vessel tortuosity and artifacts
* bifucation lesion needs complex procedure with insert two or more Drug eluting stents.
* lesion length >30mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute myocardial infarction including ST-segment elevation myocardial infarction (STEMI) or non ST-segment elevation myocardial infarction (NSTEMI) treated with PCI
Sampling Method: Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of malapposed and uncovered stent strut at 12±1 months in both DES groups | 12month
  Incidence of malapposed and uncovered stent strut measured by OCT

SECONDARY OUTCOMES:
Percent neointima cross-sectional area | 12month
  By OCT, percentage neointima cross sectional area can be obtained by dividing the neointimal area by the stent area.(neointima cross-sectional area in mm²(Quadratmillimeter)/sec)
Mean neointima thickness | 12month
  By OCT, neointima thickness can be measured as distance from the endoluminal surface of the neointima to the stent strut.(mean neointima thickness in millimeter)
Morphologic characteristics of neointima | 12month
  Morphologic characteristics of neointima measured by OCT(morphologic characteristics of neointima is one of fibrous, fibrocalcific, lipid-laden)

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Ho Hur, Postdoctoral, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- Keimyung University Dongsan Medical Center, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Qian J, Zhang YJ, Xu B, Yang YJ, Yan HB, Sun ZW, Zhao YL, Tang YD, Gao Z, Chen J, Cui JG, Mintz GS, Gao RL. Optical coherence tomography assessment of a PLGA-polymer with electro-grafting base layer versus a PLA-polymer sirolimus-eluting stent at three-month follow-up: the BuMA-OCT randomised trial. EuroIntervention. 2014 Nov;10(7):806-14. doi: 10.4244/EIJY14M07_17. PMID 25033105
- [Background] Gwon HC, Hahn JY, Park KW, Song YB, Chae IH, Lim DS, Han KR, Choi JH, Choi SH, Kang HJ, Koo BK, Ahn T, Yoon JH, Jeong MH, Hong TJ, Chung WY, Choi YJ, Hur SH, Kwon HM, Jeon DW, Kim BO, Park SH, Lee NH, Jeon HK, Jang Y, Kim HS. Six-month versus 12-month dual antiplatelet therapy after implantation of drug-eluting stents: the Efficacy of Xience/Promus Versus Cypher to Reduce Late Loss After Stenting (EXCELLENT) randomized, multicenter study. Circulation. 2012 Jan 24;125(3):505-13. doi: 10.1161/CIRCULATIONAHA.111.059022. Epub 2011 Dec 16. PMID 22179532
- [Background] Kim S, Kim JS, Shin DH, Kim BK, Ko YG, Choi D, Cho YK, Nam CW, Hur SH, Jang Y, Hong MK. Comparison of early strut coverage between zotarolimus- and everolimus-eluting stents using optical coherence tomography. Am J Cardiol. 2013 Jan 1;111(1):1-5. doi: 10.1016/j.amjcard.2012.08.037. Epub 2012 Oct 2. PMID 23040589
- [Background] Karjalainen PP, Varho V, Nammas W, Mikkelsson J, Pietila M, Ylitalo A, Airaksinen JK, Sia J, Nyman K, Biancari F, Kiviniemi T. Early neointimal coverage and vasodilator response following biodegradable polymer sirolimus-eluting vs. durable polymer zotarolimus-eluting stents in patients with acute coronary syndrome -HATTRICK-OCT trial. Circ J. 2015;79(2):360-7. doi: 10.1253/circj.CJ-14-1000. Epub 2014 Dec 15. PMID 25502167
- [Derived] Lee CH, Lee S, Hwang J, Kim IC, Cho YK, Yoon HJ, Kim H, Nam CW, Hur SH. Late stent strut apposition and coverage after drug-eluting stent implantation by optical coherence tomography in patients with acute myocardial infarction. Coron Artery Dis. 2025 Nov 1;36(7):610-617. doi: 10.1097/MCA.0000000000001536. Epub 2025 Sep 24. PMID 40421609